CLINICAL TRIAL: NCT06127875
Title: Effects of Trying to Conceive Using an Home- or Hospital-based Ovulation Monitoring on Stress
Status: Completed | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-HS-115
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-10

CONDITIONS: Fertility Issues; Stress, Psychological
Keywords: Psychological stress; Ovulation Monitoring; anxiety; depression; Sexual intercourse
MeSH Terms: conditions — Infertility; Stress, Psychological; Anxiety Disorders; Depression; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Home Ovulation Monitoring Group: timed intercourse by predicting the ovulation period or using ovulation test strips
- Hospital Ovulation Monitoring Group: timed intercourse by ultrasound ovulation monitoring

SUMMARY:
The goal of this observational study is to compare the difference of stress level and anxiety and depression between couples under home ovulation monitoring and hospital ultrasound monitoring.And whether it has a negative effect on the couple's sexual behavior.The participants were all healthy couples with fertility requirements from the reproductive Center of the First Hospital of Jilin University.The main questions it aims to answer are:

* [question1] : Does ultrasound monitoring of ovulation increase stress levels and anxiety and depression in couples trying to conceive?
* [question2] : Does ovulation monitoring affect couples' sexual function and satisfaction? Participants will be asked to fill out questionnaires three times over four menstrual cycles.

DETAILED DESCRIPTION:
The goal of this observational study is to compare the difference of stress level and anxiety and depression between couples under home ovulation monitoring and hospital ultrasound monitoring.And whether it has a negative effect on the couple's sexual behavior.The participants were all healthy couples with fertility requirements from the reproductive Center of the First Hospital of Jilin University.

Each couple needs to complete three questionnaires, one after informed consent, the second after two menstrual cycles, and the third after four menstrual cycles. If the woman becomes pregnant within 4 cycles, the investigation will be stopped.

The study was divided into two groups，home ovulation monitoring group and hospital ovulation monitoring group.The questionnaires used were the Perceived Stress Scale (PSS) , the Hospital Anxiety and Depression Scale (HADS) ,Sexual functioning was assessed with the Female Sexual Function Index (FSFI) ,the International Index of Erectile Function (IIEF) and premature ejaculation diagnostic tool（PEDT）.

ELIGIBILITY:
Inclusion Criteria:

* Normal sexual activity, no contraception for more than six months, and no ovulation monitoring in any way before Preparing for ovulation monitoring

Exclusion Criteria:

* Couples with contraindications to pregnancy The man was diagnosed with severe oligozoospermia and azoospermia

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The recruiters are all couples seeking to conceive from the Reproductive Center of a university affiliated hospita. All couples are healthy. They have normal sexual intercourse without contraception, and not pregnant for more than six months.
Sampling Method: Non-Probability Sample
Enrollment: 311 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-11-09 (Actual)

PRIMARY OUTCOMES:
Will hospital ovulation monitoring increase stress levels in couples? | A year
  The questionnaires used were the Perceived Stress Scale (PSS). The instrument uses a 5-point Likert scale rating from "0 = never" to "4=very often"for 14 items. Scores can range from 0 to 56, with higher score indicates greater psychological stress. Compare whether there are differences between hospital ovulation monitoring and home ovulation monitoring.
Will hospital ovulation monitoring increase anxiety and depression in couples? | A year
  The questionnaires used were the Hospital Anxiety and Depression Scale (HADS). Each domain has seven items with score ranges of 0 to 3, and total scores of 0 to 21. Higher scores indicate higher levels of anxiety and depression. Compare whether there are differences between hospital ovulation monitoring and home ovulation monitoring.

SECONDARY OUTCOMES:
The impact of two sets of ovulation monitoring methods on sexual function | A year
  Sexual functioning was assessed with the Female Sexual Function Index (FSFI) for female and the International Index of Erectile Function (IIEF) and premature ejaculation diagnostic tool（PEDT） for male. Compare whether there are differences between hospital ovulation monitoring and home ovulation monitoring

CONTACTS AND LOCATIONS:
Overall Officials: yang yu, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- the first hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zegers-Hochschild F, Adamson GD, Dyer S, Racowsky C, de Mouzon J, Sokol R, Rienzi L, Sunde A, Schmidt L, Cooke ID, Simpson JL, van der Poel S. The International Glossary on Infertility and Fertility Care, 2017. Fertil Steril. 2017 Sep;108(3):393-406. doi: 10.1016/j.fertnstert.2017.06.005. Epub 2017 Jul 29. PMID 28760517
- [Background] Behre HM, Kuhlage J, Gassner C, Sonntag B, Schem C, Schneider HP, Nieschlag E. Prediction of ovulation by urinary hormone measurements with the home use ClearPlan Fertility Monitor: comparison with transvaginal ultrasound scans and serum hormone measurements. Hum Reprod. 2000 Dec;15(12):2478-82. doi: 10.1093/humrep/15.12.2478. PMID 11098014
- [Background] Tiplady S, Jones G, Campbell M, Johnson S, Ledger W. Home ovulation tests and stress in women trying to conceive: a randomized controlled trial. Hum Reprod. 2013 Jan;28(1):138-51. doi: 10.1093/humrep/des372. Epub 2012 Oct 18. PMID 23081872
- [Background] Weddell S, Jones GL, Duffy S, Hogg C, Johnson S, Ledger W. Home ovulation test use and stress during subfertility evaluation: Subarm of a randomized controlled trial. Womens Health (Lond). 2019 Jan-Dec;15:1745506519838363. doi: 10.1177/1745506519838363. PMID 30924413
- [Background] Martins MV, Fernandes J, Pedro J, Barros A, Xavier P, Schmidt L, Costa ME. Effects of trying to conceive using an every-other-day strategy versus fertile window monitoring on stress: a 12-month randomized controlled trial. Hum Reprod. 2022 Nov 24;37(12):2845-2855. doi: 10.1093/humrep/deac228. PMID 36272105
- [Background] Ahn SH, Lee I, Cho S, Kim HI, Baek HW, Lee JH, Park YJ, Kim H, Yun BH, Seo SK, Park JH, Choi YS, Lee BS. Predictive Factors of Conception and the Cumulative Pregnancy Rate in Subfertile Couples Undergoing Timed Intercourse With Ultrasound. Front Endocrinol (Lausanne). 2021 Apr 15;12:650883. doi: 10.3389/fendo.2021.650883. eCollection 2021. PMID 33935968
- [Background] Gibbons T, Reavey J, Georgiou EX, Becker CM. Timed intercourse for couples trying to conceive. Cochrane Database Syst Rev. 2023 Sep 15;9(9):CD011345. doi: 10.1002/14651858.CD011345.pub3. PMID 37709293
- [Background] Song SH, Kim DS, Yoon TK, Hong JY, Shim SH. Sexual function and stress level of male partners of infertile couples during the fertile period. BJU Int. 2016 Jan;117(1):173-6. doi: 10.1111/bju.13201. Epub 2015 Jul 14. PMID 26074135
- [Derived] Xi Q, Kong Q, Lv X, Dai R, Yu Y. Impact of ejaculation frequency on semen parameters and DNA fragmentation: a cross-sectional study. Reprod Biol Endocrinol. 2025 Jul 16;23(1):100. doi: 10.1186/s12958-025-01439-3. PMID 40671092